CLINICAL TRIAL: NCT05257655
Title: MRI Observation After Ganglionic Local Opioid Analgesia at the Ganglion Cervicale Superius
Brief Title: Ganglionic Local Opioid Analgesia at the Ganglion Cervicale Superius
Acronym: GLOA-MRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Klagenfurt am Wörthersee (Other)
Collaborators: University of Klagenfurt (Other)
Responsible Party: Principal Investigator, Rudolf Likar, Prim. Univ. Prof. Dr. MSc., Klinikum Klagenfurt am Wörthersee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0815-2021
Record Dates: First submitted 2022-01-31; First posted 2022-02-25 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Trigeminal Neuralgia, Idiopathic; Postherpetic; Neuralgia, Trigeminal (Etiology); Glossopharyngeal Neuralgia; Atypical Facial Pain
Keywords: GLOA, MRI,
MeSH Terms: conditions — Trigeminal Neuralgia; Neuralgia; Glossopharyngeal Nerve Diseases

STUDY DESIGN:
Intervention Model Description: Single treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): MRI after Ganglionic Local Opioid Analgesia at the Ganglion Cervicale Superius;
  Interventions: Procedure: MRI after ganglionic local opioid analgesia (GLOA)

INTERVENTIONS:
Procedure: MRI after ganglionic local opioid analgesia (GLOA) — MRI after Ganglionic Local Opioid Analgesia at the Ganglion Cervicale Superius
  Other Names: MRI

SUMMARY:
The blockade of the superior cervical ganglion (GCS) of the sympathetic trunk is a very special form of therapy. The transoral blocking technique, also known as GLOA (ganglionic local opioid analgesia), is very suitable for achieving GCS. A total of 5 μg of sufentanil in 2 ml of sodium chlorid are applied.

Since no imaging evidence of the injected substances has been published for a GLOA in a living person, it is planned to carry out an MRI examination immediately after the ganglionic local opioid analgesia in order to show the spread and distribution pattern of the injected substance. It is also planed to show a correlation of the spread of the injected substance with the efficacy of the intervention.

To determine the interrater reliability, the GLOA is carried out alternately by 2 different examiners and the existing MRI images of the GLOA are assessed by an radiologist and anatomist in a blinded manner.

In a follow-up after 1 and 3 months, the questionnaires and pain scores are evaluated again.

DETAILED DESCRIPTION:
The blockade of the superior cervical ganglion (GCS) of the sympathetic trunk is a very special form of therapy. It is successfully used for numerous, often protracted diseases that severely impair the patient's quality of life, such as idiopathic facial pain syndromes or trigeminal neuralgia. The transoral blocking technique, also known as GLOA (ganglionic local opioid analgesia), is very suitable for achieving GCS. With this technique, a Sprotte cannula is inserted into the pharyngeal recess (Rosenmueller) located behind the palatopharyngeal arch and pierced through the pharyngeal wall into the parapharyngeal space. A total of 5 μg of sufentanil in 2 ml of sodium chlorid are applied.

Since no imaging evidence of the injected substances has been published for a GLOA in a living person, it is planned to carry out an MRI examination immediately after the ganglionic local opioid analgesia in order to show the spread and distribution pattern of the injected substance. It is also planed to show a correlation of the spread of the injected substance with the efficacy of the intervention. For this, different questionnaires (NRS, quality of life, sleep quality, patient satisfaction) are carried out before and after the intervention.

To determine the interrater reliability, the GLOA is carried out by 2 different examiners and the existing MRI images of the GLOA are assessed by an radiologist and anatomist in a blinded manner.

In a follow-up after 1 and 3 months, the questionnaires and pain scores are evaluated again.

ELIGIBILITY:
Inclusion Criteria:

* Trigeminal neuralgia
* Postherpetic neuralgia
* Glossopharyngeal neuralgia
* Atypical facial pain

Exclusion Criteria:

* psychosis
* language barrier
* Pregnant and breastfeeding women
* Seizure disorders (epilepsy)
* Increased risk of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Distribution of the injected fluid in the area of the superior cervical ganglion | immediately after the intervention
  MRI verified distribution of the injected fluid in the area of the superior cervical ganglion

SECONDARY OUTCOMES:
Quality of life questionnaire | Before first and after last GLOA. After 1 and 3 month (follow up)
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state (https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/)
Pain assessed by NRS | baseline, immediately after intervention, After 1 and 3 month (follow up)
  Present pain intensity on a 0-10 Numerical Rating Scale (NRS) with 0 corresponding to "no pain" and 10 to "the worst pain imaginable
Patient satisfaction assessed by satisfaction questionaire | Before first and after last GLOA. After 1 and 3 month (follow up)
  ZUF-8 is a measuring instrument for the global, one-dimensional recording of patient satisfaction. It is the German-language adaptation of the American CSQ-8 by Attkisson & Zwick (1982). General satisfaction ("general satisfaction") with aspects of the clinic or the treatment received is recorded using eight items. ZUF-8 is particularly suitable for an economical screening of patient satisfaction.
Sleep quality assessed by sleep quality questionnaire | Before first and after last GLOA. After 1 and 3 month (follow up)
  To record the sleep quality the questionnaire on sleep quality is carried out (PSQI)
Efficacy prediction based on MRI verified fluid spread | immediately after the intervention
  Efficacy prediction based on the MRI verified fluid spread in millimeter in the area of the superior cervical ganglion

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Likar, Prof., Principal Investigator — Klinikum Klagenfurt am Wörthersee
Locations (1):
- Klinikum Klagenfurt am Wörthersee, Klagenfurt, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feigl G, Rosmarin W, Likar R. [Block of the superior cervical ganglion of the Truncus sympathicus. Why it often is not possible!]. Schmerz. 2006 Aug;20(4):277-80, 282-4. doi: 10.1007/s00482-005-0435-6. German. PMID 16142462
- [Background] Spacek A, Bohm D, Kress HG. Ganglionic local opioid analgesia for refractory trigeminal neuralgia. Lancet. 1997 May 24;349(9064):1521. doi: 10.1016/S0140-6736(05)62101-0. No abstract available. PMID 9167469
- [Derived] Neuwersch-Sommeregger S, Kostenberger M, Sandner-Kiesling A, Furstner M, Igerc I, Trummer B, Wuntschek J, Pipam W, Stettner H, Likar R, Feigl G. Ganglionic Local Opioid Analgesia at the Superior Cervical Ganglion: MRI-Verified Solution Spread. Pain Ther. 2024 Jun;13(3):663-678. doi: 10.1007/s40122-024-00596-4. Epub 2024 Apr 25. PMID 38662320